CLINICAL TRIAL: NCT04222075
Title: Identification of the Impact of Acute Pancreatitis on Quality of Life in Discharged Chinese Patients: a One-year Follow-up Study
Brief Title: Identification of the Impact of Acute Pancreatitis on Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, DONG WU, Associate Professor of Gastroenterology, Peking Union Medical College Hospital
Other Study IDs: WD-2018APQOL
Record Dates: First submitted 2019-12-11; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Acute Pancreatitis; Quality of Life
Keywords: Acute Pancreatitis; Quality of Life
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Pancreatitis: Patients after acute pancreatitis

SUMMARY:
In abdomen, the pancreas as a gland is involved in the digestive and endocrine system by secreting digestive enzymes and insulin. Acute pancreatitis (AP) is a common inflammatory condition of the pancreas with symptoms of sudden abdominal pain and high temperature which may develop to severe complications in some patients. The incidence of AP was roughly 33.74 cases per 100, 000 person-years around the world but varies in different regions which America has the highest incidence of 58.20 cases per 100 000 person-years. There are very few studies published on AP in China, while Japanese national survey in 2011 estimated an incidence rate of 49.4 per 100,000 population and a study in Taiwan showed an annual average incidence of 36.9 per 100,000 persons with a slight change over ten years.

In most cases, patient with AP will start to recover within a week, but the patient quality of life (QoL) is still a big concern for disease management. It quantitatively measures the physical, mental and social wellbeing of individuals or their life satisfaction by questionnaires or surveys. Although very few studies have demonstrated the effect of AP on patient QoL, there is accumulating evidence to show its importance. Some studies reported no differences in QoL between AP patients and age-matched healthy people, whereas others showed QoL was significantly impaired due to AP. A large population-based follow-up study is needed to evaluate the impact of acute pancreatitis on quality of life. In addition, as the population investigated in most research was European based, the QoL evaluation of patients after AP among the Chinese population is also essential.

ELIGIBILITY:
Inclusion Criteria:

* Acute pancreatitis.
* Must be able to response an online survey.

Exclusion Criteria:

• N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to Peking Union Medical College Hospital with a diagnosis of acute pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-26 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life of patients after acute pancreatitis will be assessed by EuroQol five-dimension three-level questionnaire (One-month follow-up after discharge) | 1 month
  Onemonth follow-up after discharge: Quality of life of patients after acute pancreatitis will be assessed by EuroQol five-dimension three-level (EQ-5D-3L) questionnaire, which essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems (1), some problems (2), and extreme problems (3). As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions). Chinese Time-Trade Off value sets will be adopted to transform the descriptive system into health value (-0.149 to 1). The higher health value indicates the better health status.
Quality of life of patients after acute pancreatitis will be assessed by EuroQol five-dimension three-level questionnaire (Three-month follow-up after discharge) | 3 months
  Three-month follow-up after discharge: Quality of life of patients after acute pancreatitis will be assessed by EuroQol five-dimension three-level (EQ-5D-3L) questionnaire, which essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems (1), some problems (2), and extreme problems (3). As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions). Chinese Time-Trade Off value sets will be adopted to transform the descriptive system into health value (-0.149 to 1). The higher health value indicates the better health status.
Quality of life of patients after acute pancreatitis will be assessed by EuroQol five-dimension three-level questionnaire (Six-month follow-up after discharge) | 6 months
  Six-month follow-up after discharge: Quality of life of patients after acute pancreatitis will be assessed by EuroQol five-dimension three-level (EQ-5D-3L) questionnaire, which essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems (1), some problems (2), and extreme problems (3). As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions). Chinese Time-Trade Off value sets will be adopted to transform the descriptive system into health value (-0.149 to 1). The higher health value indicates the better health status.
Quality of life of patients after acute pancreatitis will be assessed by EuroQol five-dimension three-level questionnaire (Twelve-month follow-up after discharge) | 12 months
  Twelve-month follow-up after discharge: Quality of life of patients after acute pancreatitis will be assessed by EuroQol five-dimension three-level (EQ-5D-3L) questionnaire, which essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems (1), some problems (2), and extreme problems (3). As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions). Chinese Time-Trade Off value sets will be adopted to transform the descriptive system into health value (-0.149 to 1). The higher health value indicates the better health status.

SECONDARY OUTCOMES:
Quality of life of patients after acute pancreatitis will be assessed by 36-Item Short-form health survey (One-month follow-up after discharge) | 1 month
  One-month follow-up after discharge: Quality of life of patients after acute pancreatitis will be assessed by 36-Item Short-form health survey (SF-36), which is a 36-item, patient-reported survey of patient health. It consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Quality of life of patients after acute pancreatitis will be assessed by 36-Item Short-form health survey (Three-month follow-up after discharge) | 3 months
  Three-month follow-up after discharge: Quality of life of patients after acute pancreatitis will be assessed by 36-Item Short-form health survey (SF-36), which is a 36-item, patient-reported survey of patient health. It consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Quality of life of patients after acute pancreatitis will be assessed by 36-Item Short-form health survey (Six-month follow-up after discharge) | 6 months
  Six-month follow-up after discharge: Quality of life of patients after acute pancreatitis will be assessed by 36-Item Short-form health survey (SF-36), which is a 36-item, patient-reported survey of patient health. It consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Quality of life of patients after acute pancreatitis will be assessed by 36-Item Short-form health survey (Twelve-month follow-up after discharge) | 12 months
  Twelve-month follow-up after discharge: Quality of life of patients after acute pancreatitis will be assessed by 36-Item Short-form health survey (SF-36), which is a 36-item, patient-reported survey of patient health. It consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.

CONTACTS AND LOCATIONS:
Overall Officials: DONG WU, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Pendharkar SA, Salt K, Plank LD, Windsor JA, Petrov MS. Quality of life after acute pancreatitis: a systematic review and meta-analysis. Pancreas. 2014 Nov;43(8):1194-200. doi: 10.1097/MPA.0000000000000189. PMID 25333403
- [Background] Machicado JD, Gougol A, Stello K, Tang G, Park Y, Slivka A, Whitcomb DC, Yadav D, Papachristou GI. Acute Pancreatitis Has a Long-term Deleterious Effect on Physical Health Related Quality of Life. Clin Gastroenterol Hepatol. 2017 Sep;15(9):1435-1443.e2. doi: 10.1016/j.cgh.2017.05.037. Epub 2017 Jun 1. PMID 28579182
- [Derived] Ding H, Dai J, Lin J, Gong L, Sun H, Song K, Xie F, Wu D. A 12-month follow-up study of discharged patients with acute pancreatitis: An acute condition with prolonged sequela. Chin Med J (Engl). 2024 Jan 20;137(2):250-252. doi: 10.1097/CM9.0000000000002847. Epub 2023 Sep 5. No abstract available. PMID 37668021